CLINICAL TRIAL: NCT04801810
Title: Effects of Daily Low Oxygen Exposure on Weight Status, Body Composition, and Metabolic Health
Brief Title: Daily Low Oxygen Exposure and Weight Status
Acronym: LOWS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was registered in conjunction with a submitted R01. To address reviewer comments, the study was changed substantially for resubmission. A new study has been registered (NCT05289310) that aligns with the funded R01.
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Claire E. Berryman, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000334
Record Dates: First submitted 2021-03-07; First posted 2021-03-17 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Overweight and Obesity
Keywords: Body weight; Normobaric hypoxia; Overwieght and obesity; Negative energy balance; Energy expenditure; Energy intake
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric hypoxia (NH) (Experimental): 8 weeks of overnight exposure (8 hrs/night) to NH conditions (~15% oxygen; achieved with nitrogen dilution, equivalent to ~8500 feet elevation) using a commercially available tent and generator system (Hypoxico, Inc., New York, NY).
  Interventions: Other: Normobaric hypoxia
- Normobaric normoxia (NN) (Sham Comparator): 8 weeks of overnight exposure (8 hrs/night) to NN conditions (~21% oxygen; sea level) using a commercially available tent and generator system (Hypoxico, Inc., New York, NY).
  Interventions: Other: Normobaric normoxia

INTERVENTIONS:
Other: Normobaric hypoxia — Low oxygen exposure to mimic ~8500 feet elevation (experimental).
  Arms: Normobaric hypoxia (NH)
Other: Normobaric normoxia — Normal oxygen exposure to mimic sea level conditions (sham comparator).
  Arms: Normobaric normoxia (NN)

SUMMARY:
The objective of this single-blind, parallel-arm, randomized clinical trial is to evaluate changes in body weight and composition, assess determinants of energy balance, and measure modulators of energy intake and expenditure, following 8 wk of calorie restriction (CR, -500 kcal/d) in combination with either overnight exposure (8 h/night) to normobaric hypoxia (NH; 15% oxygen, ~8500 ft elevation) or normoxia (NN; 21% oxygen, sea level), using a commercially available, in-home tent system, in adults who are overweight or obese.

DETAILED DESCRIPTION:
The current research study will evaluate changes in body weight and composition, assess determinants of energy balance, and measure modulators of energy intake and expenditure, following 8 wk of calorie restriction (CR, -500 kcal/d) in combination with either overnight exposure to normobaric hypoxia (NH) or normoxia (NN). Participants will be instructed to follow their normal diet but with a 500 kcal/day deficit as advised by a Registered Dietitian. Participants will spend 8 hours/night in a tent, set-up around their bed, in their home, for 8 weeks. Participants sleeping in the hypoxic tent (Hypoxico Inc., New York, NY, commercially available tents: https://hypoxico.com/) will breath ~15% oxygen (achieved with nitrogen dilution, equivalent to ~8500 ft elevation), whereas those in the control tent (Hypoxico Inc.) will breath ~21% oxygen (achieved with nitrogen dilution, equivalent to sea level elevation). Trained research staff will set-up the hypoxic or control tent system in each participant's home on day 0 and will visit the participant's home on days 1, 2, and 3 to check and/or adjust the tent settings. After day 3, research staff will visit the participant's home weekly to check and/or adjust the tent settings. participants will be weighed each morning following an overnight fast and morning void. Participants will come to the laboratory on two separate days for baseline testing (days -1 and 0) and again on two separate days at the end of the study (days 55 and 56) for endpoint testing.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20 - 50 years
* Overweight or obese (BMI between 27.5-34.9 kg/m2)
* Born at altitudes less than 2,100 meters (~7,000 feet)
* Currently residing in Tallahassee, Florida, or the surrounding area
* Not taking any medication(s) that interfere with metabolism or oxygen delivery/transport for 4 weeks prior to and throughout the entire study (e.g., includes sedatives, sleeping aids, tranquilizers, and/or any medication that depresses ventilation, diuretics, alpha, and beta-blockers).
* Willing to refrain from smoking, vaping, chewing tobacco, and dietary supplement use throughout the entire study
* Willing to have a hypoxic tent set-up in their home and spend 8 consecutive hours per night in the tent for 8 weeks
* Lives with a family member, partner/spouse, or roommate who can hear and respond in the unlikely event that the blood oxygen, air oxygen, or air carbon dioxide monitoring alarm would sound.

Exclusion Criteria:

* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for five days or more within the last 2 months
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders, and any condition that interferes with metabolism or oxygen delivery/transport (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Evidence of apnea or other sleeping disorders
* Evidence of prior high-altitude pulmonary edema (HAPE) or high-altitude cerebral edema (HACE) diagnosis
* Diagnosis or family history of sickle cell anemia/trait
* Hematocrit <42% for males, <36% for females
* Hemoglobin <13 g/dL for males, <12 g/dL for females
* Blood donation within 8 weeks of beginning the study
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Allergies or intolerance to foods included in the standardized and ad libitum meal tests (e.g., lactose intolerance/milk allergy)
* Women who are pregnant, lactating, planning to become pregnant, or who have had an irregular menstrual cycle in the past 6 mo.
* Weight gain or loss > 10% of body weight during the past 6 months
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight | 8 weeks (56 days)
  Body weight will be measured during baseline (days -7 to 0) and each morning during the study (days 1 to 56) following an overnight fast and morning void, using a calibrated digital scale provided to participants to use at home (A&D Medical wireless weight scale UC-352BLE, San Jose, CA). Percent change in body weight will be calculated as:
  [Body weight - baseline body weight (average of days -7 to 0)]/ baseline body weight * 100

SECONDARY OUTCOMES:
Percent change in body weight | 4 weeks after intervention ends
  Body weight also will be measured 4 weeks after the study intervention ends to assess whether weight loss is sustained.
4-compartment body composition using DEXA and deuterium dilution | Days -1 and 55
  Body composition will be determined following a 12 hour fast and morning void on day -1 and 55 using dual energy x-ray absorptiometry (DEXA, Discovery W, Hologic Inc., Bedford, MA or equivalent). The volunteer will remove all metal-containing objects from their body, lay face-up on the DEXA densitometer table in light clothing (t-shirt, shorts, socks), and be asked to remain motionless for the 8-10 min scan. A scanner emitting low energy x-rays and a detector will pass over the participant. These data will be used to calculate total body mass, fat-free mass, fat mass, and bone mass. Total body water will be measured following a 12 hour fast and 1 hour without water intake using the deuterium dilution method on days -1 and 55.
Resting metabolic rate | Days 0 and 56
  Resting metabolic rate will be measured with open circuit, indirect calorimetry (ParvoMedics TrueOne 2400 metabolic cart, Sandy, UT) in the morning, upon arrival to the lab on days 0 and 56.
Resting substrate oxidation | Days 0 and 56
  Resting substrate oxidation will be measured with open circuit, indirect calorimetry (ParvoMedics TrueOne 2400 metabolic cart, Sandy, UT) in the morning, upon arrival to the lab on days 0 and 56.
Total daily energy intake | Weeks -1, 1, 2, 4, 6, and 8
  Participants will complete 3 dietary records (2 week days, 1 weekend day) prior to the in-person baseline visit and during weeks 1, 2, 4, 6, and 8 of the study using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool. This web-based tool was developed by the National Cancer Institute: https://epi.grants.cancer.gov/asa24/.
Total daily macronutrient intake | Weeks -1, 1, 2, 4, 6, and 8
  Participants will complete 3 dietary records (2 week days, 1 weekend day) prior to the in-person baseline visit and during weeks 1, 2, 4, 6, and 8 of the study using the Automated Self-Administered 24-Hour (ASA24®) Dietary Assessment Tool. This web-based tool was developed by the National Cancer Institute: https://epi.grants.cancer.gov/asa24/.
Ad libitum energy intake | Days 0 and 56
  Ad libitum energy intake will be assessed by measuring total energy intake during an ad libitum buffet-style meal provided to participants on days 0 and 56.
Food preferences | Days 0 and 56
  Food preferences will be assessed by measuring macronutrient intake during an ad libitum buffet-style meal provided to participants on days 0 and 56.
Heart rate variability | Days 0 and 56
  A 3-lead electrocardiogram will be conducted on days 0 and 56 to assess heart rate variability. Participants will have electrode patches placed on their chest to measure the electrical activity of the heart.
Urinary epinephrine | Days -1, 13, and 55
  On days -1, 13, and 55 urine will be collected during the overnight time period. Participants will void their bladder before entering the tent in the evening (they will not collect this portion). Participants will collect any urine produced throughout the night and will collect one final time in the morning after exiting the tent. Epinephrine concentrations in the urine samples will be measured.
Urinary norepinephrine | Days -1, 13, and 55
  On days -1, 13, and 55 urine will be collected during the overnight time period. Participants will void their bladder before entering the tent in the evening (they will not collect this portion). Participants will collect any urine produced throughout the night and will collect one final time in the morning after exiting the tent. Norepinephrine concentrations in the urine samples will be measured.
Urinary dopamine | Days -1, 13, and 55
  On days -1, 13, and 55 urine will be collected during the overnight time period. Participants will void their bladder before entering the tent in the evening (they will not collect this portion). Participants will collect any urine produced throughout the night and will collect one final time in the morning after exiting the tent. Dopamine concentrations in the urine samples will be measured.
Plasma glucose concentrations | Days 0 and 56
  A 75-g oral glucose tolerance test (OGTT) will be conducted on days 0 and 56. A venous catheter will be placed and blood samples obtained at -5, 30, 60, 90, and 120 min during the OGTT for measurements of plasma glucose and insulin concentration. Insulin sensitivity will be determined by using the whole-body insulin sensitivity index (WBISI), also known as the Matsuda Index.
Plasma insulin concentrations | Days 0 and 56
  A 75-g oral glucose tolerance test (OGTT) will be conducted on days 0 and 56. A venous catheter will be placed and blood samples obtained at -5, 30, 60, 90, and 120 min during the OGTT for measurements of plasma glucose and insulin concentration. Insulin sensitivity will be determined by using the whole-body insulin sensitivity index (WBISI), also known as the Matsuda Index.
Whole-body insulin sensitivity index | Days 0 and 56
  A 75-g oral glucose tolerance test (OGTT) will be conducted on days 0 and 56. A venous catheter will be placed and blood samples obtained at -5, 30, 60, 90, and 120 min during the OGTT for measurements of plasma glucose and insulin concentration. Insulin sensitivity will be determined by using the whole-body insulin sensitivity index (WBISI), also known as the Matsuda Index.
Thermic effect of glucose | Days 0 and 56
  The thermic effect of glucose will be measured on study days 0 and 56 with open circuit, indirect calorimetry (2400 TrueOne, Parvo Medics) using established protocols. Resting metabolic rate measurements will be taken prior to glucose administration in a thermo-neutral room while the participant is in the supine position (as described above). During the oral glucose tolerance test the thermic effect of glucose will be measured in 15 min increments for 2 hours (15-30, 45-60, 75-90, and 105-120 minutes).
Subjective appetite measures | Days 0 and 56
  Subjective appetite will be measured on study days 0 and 56. Subjectively rated appetite will be assessed immediately before the oral glucose tolerance test (OGTT) and at 15, 30, 45, 60, 90, and 120 minutes after beginning the OGTT using 100 mm visual analog scales to rate fullness, hunger, desire to eat, and prospective food consumption. Composite satiety score will be calculated from the individual appetite scores using the equation: CSS = (fullness + (100 - Desire to eat) + (100 - Hunger) + (100 - Prospective food consumption) / 4.
Prevalence of acute mountain sickness | Days 0-7, 14, 21, 28, 35, 42, and 56
  The prevalence and severity of acute mountain sickness (AMS) will be determined from information gathered using the shortened version of the Environmental Symptoms Questionnaire (ESQ) (5 min; 26 questions total). The minimum score is 0 and the maximum score is 5. A lower score indicates fewer AMS symptoms. At completion, oxygen saturation will be determined using finger pulse oximetry (PalmSAT® 2500A, Nonin Medical, Inc., Plymouth, MN). AMS and oxygen saturation measurements will be taken in the morning on days 0-7, 14, 21, 28, 35, 42, and 56.
Continuous overnight oxygen saturation | 8 weeks (56 days)
  Oxygen saturation will be measured continuously overnight (8 h/night) using a finger pulse oximeter (PalmSAT® 2500, Nonin Medical, Inc., Plymouth, MN) during 8 weeks of overnight exposure to NH or NN.
Sleep quality | Days 0-7, 14, 28, 35, 42, and 56
  The Pittsburgh Sleep Quality Index (PSQI; 5 minutes, 18 questions) will be used to examine volunteer sleep quality on days 0-7, 14, 28, 35, 42, and 56. The minimum score is 0 and the maximum score is 21. Lower scores indicate better sleep quality.
24-hour continuous glucose concentrations | Days -7 to 0, 1 to 14, and 42 to 56
  A continuous glucose monitor (Freestyle Libre Pro) will be inserted into the subcutaneous adipose tissue behind the arm and will be used to collect and assess 24-hour glucose concentrations during baseline (day -7 to day 0), days 1-14, and days 42-56.
24-hour glucose variability | Days -7 to 0, 1 to 14, and 42 to 56
  A continuous glucose monitor (Freestyle Libre Pro) will be inserted into the subcutaneous adipose tissue behind the arm and will be used to collect and assess 24-hour glucose concentrations during baseline (day -7 to day 0), days 1-14, and days 42-56.
Blood volume | Days -1 and 55
  Blood volume will be determined using the optimized carbon monoxide rebreathing method on days -1 and 55. In this method, a capillary blood sample is taken, and basal carboxyhemoglobin concentrations will be determined using a blood gas analyzer. Carbon monoxide is then inhaled via a spirometer (SpiCo, Blood Tec.) for 2 minutes. Seven minutes after inhaling the carbon monoxide bolus, a second capillary blood sample is taken to determine the increase in carboxyhemoglobin concentration. The change in percentage of carboxyhemoglobin between the basal and second measurements can be used to calculate hemoglobin mass and blood volume.
Fasting measures of iron status | Days 0 and 56
  Serum iron, total iron binding capacity, soluble transferrin receptor, hepcidin, hemoglobin, hematocrit, ferritin, erythroferrone, and erythropoietin will be measured in fasting blood samples collected on days 0 and 56.
Psychosocial Factors | Days -1, 14, and 55
  The Positive and Negative Affect Schedule, Cohen Perceived Stress Scale, Big Five Inventory-2, Delay Discounting questionnaire, Palatable Eating Motives Scale, and the Generalized Self-Efficacy scale will be administered on days -1, 14, and 55.
Fasting blood pressure | Days 0 and 56
  Fasting blood pressure will be measured on days 0 and 56 using an automated blood pressure cuff. All blood pressure readings will be taken on the right arm, and participants will be in a seated position, after resting for at least 5 minutes. Blood pressure will be measured in triplicate.

CONTACTS AND LOCATIONS:
Overall Officials: Claire E Berryman, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No